CLINICAL TRIAL: NCT00720096
Title: A Pilot Prospective Trial Of Genomic Directed Salvage Chemotherapy With Either Liposomal Doxorubicin Or Topotecan In Recurrent Or Persistent Ovarian Cancer Within 12 Months Of Platinum-Based Chemotherapy
Brief Title: Genomic Directed Salvage Chemotherapy With Either Liposomal Doxorubicin Or Topotecan
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funds for this project have been spent, and it is thereby terminated.
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-15042; NFGC 12-12990-01-29 (Other: NFGC)
Record Dates: First submitted 2008-07-21; First posted 2008-07-22 (Estimated); Results first posted 2011-02-16 (Estimated); Last update posted 2018-01-02 (Actual); Status verified 2017-12

CONDITIONS: Ovarian Cancer
Keywords: Persistent Ovarian Cancer; Genomic directed salvage chemotherapy; Genomic Microarray
MeSH Terms: conditions — Ovarian Neoplasms | interventions — liposomal doxorubicin; Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Liposomal Doxorubicin (Experimental): Liposomal Doxorubicin - Chemotherapy single agent systemic.
  Interventions: Drug: Liposomal Doxorubicin
- Topotecan (Experimental): Topotecan - Chemotherapy single agent systemic.
  Interventions: Drug: Topotecan

INTERVENTIONS:
Drug: Liposomal Doxorubicin — Liposomal Doxorubicin 40 mg/m2 q 28 days
  Other Names: Doxil
  Arms: Liposomal Doxorubicin
Drug: Topotecan — 1. Topotecan (daily x 5 days of a 21 day cycle)
  2. Per amendment #15: Topotecan (days 1, 8, 15 of a 28 day cycle)
  Other Names: Hycamtin
  Arms: Topotecan

SUMMARY:
This pilot study will help us to determine the success of using a special technique called microarray technology to examine cancer genes in order to predict how individual women will respond to one of two therapies, liposomal doxorubicin or topotecan, and which will be more effective in treating ovarian cancer that has returned (recurrent ovarian cancer). We believe that this study may lead to a means by which microarray technology can predict the most effective treatment decision, based on the genetic characteristics of her tumor tissue, for a woman with recurrent ovarian cancer.

Another purpose of this study is to determine how quickly a woman with recurrent ovarian cancer will respond to treatment (treatment response rate) and to evaluate the accuracy of the genomic predictions.

Recent data suggest that microarray technology can predict a patient's response to chemotherapy; this has not yet been proven in a forward-looking study which is why we are conducting this research.

DETAILED DESCRIPTION:
Patients who take part in the study will have an initial visit and undergo a CT guided core biopsy. Using tissue from a CT guided core biopsy, microarray analysis will be performed to help predict which of the two drugs appears to be better suited to individual genomic factors. The results will result in being assigned to treatment with either liposomal doxorubicin or topotecan.

Patients who receive liposomal doxorubicin - IV chemotherapeutic treatment will occur 3 times, 28 days apart, weeks 1,5,and 9. At each of these visits patients will be evaluated and have blood work to check their liver tests and electrolytes. Every 8 weeks patients will have a radiologic evaluation of their tumor.

Patients who receive topotecan - IV chemotherapeutic treatment will occur 4 times, 21 days apart, weeks 1,4,7, and 10. At each of these visits patients will be evaluated and have blood work to check levels of liver tests and electrolytes. Every 8 weeks patients will have a radiologic evaluation of their tumor.

ELIGIBILITY:
Inclusion Criteria:

* Must have history of histologically or cytologically confirmed epithelial ovarian cancer with recurrence.
* Must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >20 mm with conventional techniques or as >10 mm with spiral computed tomography CT) scan.
* May have had only 2 prior chemotherapy regimens, with at least one regimen containing platinum, and disease recurrence or progression occurring between 0 to 12 months (1 to 365 days)from the platinum-containing regimen. Patients who have been treated with consolidation treatment are allowed and the consolidation will not be considered a separate regimen. Hormonal therapy and immunotherapy will not be considered a prior chemotherapy regimen. Hormonal therapies given to treat the patient's cancer should be stopped at least 30 days prior to dosing on this trial. Typical low-dose hormone replacement therapy to treat postmenopausal symptoms may be continued at the treating physician's discretion.
* Life expectancy >6 months.
* ECOG performance status 2 or less (Karnofsky 60%).
* Must have normal organ and marrow function as defined below:

  * leukocytes 3,000/microL
  * absolute neutrophil count 1,500/ microL
  * platelets 100,000/microL
  * total bilirubin ≤1.5 X institutional upper limit of normal(ULN) aspartate aminotransferase [AST(SGOT)]/alanine aminotransferase [ALT(SGPT)] ≤2.5 X ULN creatinine within normal institutional limits OR creatinine clearance 60mL/min/1.73m2 for patients with creatinine levels above institutional normal
* Ability to understand and willingness to sign a written informed consent document
* Measurable disease on CT must be considered amenable to biopsy by Core methods (core biopsy may be radiographically or non-radiographically performed). Potential ability to obtain core material must be reviewed by Principal Investigator (PI) and/or his designates prior to enrollment.
* Must consent to biopsy as part of enrolling into trial.
* Patients with reproductive potential must use an adequate contraceptive method (e.g. abstinence, intrauterine device, oral contraceptives, barrier device with spermicide or surgical sterilization) during treatment and for three months after completing treatment.
* Must have a Multiple Gated Acquisition (MUGA) scan or 2-d echocardiogram indicating an ejection fraction of > 50% or institutional standards within 42 days prior to first dose of study drug. The method used at baseline must be used for later monitoring.

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not version 13, 01/10/08 MCC 15042 16 recovered from adverse events due to agents administered more than 4 weeks earlier.
* May not be receiving any other investigational agents concurrently.
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to liposomal doxorubicin or topotecan.
* Myocardial infarction within 6 months. History of cardiac disease, with New York Heart Association Class II or greater, or clinical evidence of congestive heart failure.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Women who are pregnant.
* Women who are breastfeeding should discontinue breastfeeding.
* Human Immunodeficiency Virus (HIV)-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions and increased toxicity.
* Patients may have had no other malignancies in the prior 5 years other than non-metastatic, locally-controlled, non-melanomatous cutaneous cancers.
* Patients who have received radiation to more than 25% of marrow-bearing areas.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2008-07; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert M. Wenham, M.D., M.S., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Liposomal Doxorubicin | Topotecan
Started | 2 | 2
Completed | 2 | 0
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liposomal Doxorubicin | Topotecan | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Assess Feasibility
Description: Number of patients meeting 3 week feasibility window which was set as the benchmark.
Time Frame: 1 year, 2 months
Population: Patients whose information for treatment was available within the 3 week feasibility window which was set as the benchmark.
Measure: Number; unit: Participants
Arm/Group | Liposomal Doxorubicin | Topotecan
Number analyzed (Participants) | 2 | 2
Participants | 2 | 2

2. Primary Outcome: Interpret Genomic Array
Description: Number of patients with biopsiable tumor in sufficient quantity and quality that will result in an interpretable genomic array.
Time Frame: 1 year, 2 months
Population: All patients enrolled 4/4 had biopsiable tumor and sufficient quantity and quality.
Measure: Number; unit: Participants
Arm/Group | Liposomal Doxorubicin | Topotecan
Number analyzed (Participants) | 2 | 2
Participants
  Biopsiable tumor: sufficient quantity and quality | 2 | 2
  Interpretable data | 2 | 1

3. Secondary Outcome: Response Rate
Description: Determine response rate of array directed chemotherapy (as defined as the proportion of patients achieving complete or partial responses with a predictive score >/= 0.5 for either chemotherapy). As well as evaluate the accuracy of the chemosensitivity profiles for differentiating doxorubicin and topotecan responsive cancers. Due to the limited sample size the interpretation is limited. Results data for this outcome is not posted.
Time Frame: 1 year, 2 months
Population: Data was not collected for this Pilot study, due to small sample size and early termination.
Arm/Group | Liposomal Doxorubicin | Topotecan
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year, 2 months
Arm/Group | Liposomal Doxorubicin | Topotecan
Serious Adverse Events (participants affected / at risk) | 1/2 | 1/2
Other Adverse Events (participants affected / at risk) | 2/2 | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liposomal Doxorubicin (N=2) | Topotecan (N=2)
Hospital Admission (Reproductive system and breast disorders) | 1 (1) | 0 (0) — Pegylated Liposomal Doxorubicin (PLD) Arm Patient - patient had an SAE of hospital admission for observation due to tumor debulking done of a vaginal lesion that was deemed unrelated.
Fever combined with Anemia (General disorders) | 0 (0) | 1 (1) — Topotecan Arm Patient - patient had a hospitalization for Grade 3 neutropenic fever Grade 3 anemia deemed related to Topotecan.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liposomal Doxorubicin (N=2) | Topotecan (N=2)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Dizziness (General disorders) | 0 (0) | 1 (2)
Fatigue (General disorders) | 1 (1) | 1 (1)
Headache (General disorders) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Ant bite with infection (Infections and infestations) | 1 (1) | 0 (0)
Blister on left toe (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Blister on right toes (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Blister on right toe (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Blister on small toe left (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0)
Hand foot reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hand foot syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Increased creatinine (Renal and urinary disorders) | 0 (0) | 1 (1)
Infection in blood (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Rash (chest) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Shortage of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Syncope (General disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to limited sample size, we were unable to make definitive conclusions in this trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No